CLINICAL TRIAL: NCT04564807
Title: Testing an Online Insomnia Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Weafer (Other)
Responsible Party: Sponsor-Investigator, Jessica Weafer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60446; 1013179870 (Other Grant/Funding Number: SUPRA)
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Use Disorder; Insomnia
Keywords: sleep; cognitive behavioral therapy; CBT; electronic; alcohol; non-pharmacological
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Insomnia Education Program (Active Comparator): Adult heavy drinkers with insomnia.
  Interventions: Behavioral: Web-Based Insomnia Education Program
- SHUTi Intervention (Experimental): Adult heavy drinkers with insomnia.
  Interventions: Behavioral: SHUTi Intervention

INTERVENTIONS:
Behavioral: Web-Based Insomnia Education Program — Participants will be given access to a web-based program on sleep education to read at their own pace during the 9-week intervention period. The program content overlaps with SHUTi on the following topics: insomnia symptoms, impacts, and causes, basic sleep improvement strategies, and when to see a doctor. The information is akin to that found on WebMD or National Sleep Foundation website. Unlike the SHUTi program, the information is fixed, accessible immediately (no week-to-week information "unlocking") and there are no customized bedtime or wake-time suggestions based on sleep diary data.
  Arms: Web-Based Insomnia Education Program
Behavioral: SHUTi Intervention — Sleep Healthy Using the Internet (SHUTi) is a well-validated version of e-CBT-I comprised of 6 weekly educational modules and daily sleep diaries. Participants will have 9 weeks to complete 6 once-weekly educational "cores." Cores consist of: insomnia overview, sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention, and last approximately 45 minutes each. Participants will receive weekly objectives, as well as review and feedback on the previous core's assignments and sleep diary data, new material, assignments, and a summary. These features are supplemented with interactive features (i.e., personalized goal-setting, video vignettes). Participants receive daily emails prompting them to complete the 11-item sleep and alcohol use diary daily during the intervention.
  Arms: SHUTi Intervention

SUMMARY:
The objective of this trial is to determine the effectiveness of an electronic cognitive behavioral therapy for insomnia (e-CBT-I) module in improving sleep and reducing alcohol use among heavy drinkers with insomnia. Specifically, it will test the effectiveness of Sleep Healthy Using the Internet (SHUTi), a well-validated version of e-CBT-I comprised of 6 weekly educational modules and daily sleep diaries. The rationale for this mixed methods proposal is that effective, nonpharmacologic treatments are necessary to stem the highly comorbid public health problems of alcohol use disorder (AUD) and insomnia. If successful, SHUTi will represent a novel and easily accessible intervention for reducing alcohol intake among high-risk heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

* engage in weekly alcohol binge episodes
* moderate to severe insomnia

Exclusion Criteria:

* history of severe alcohol or other substance use disorder
* obstructive sleep apnea
* schizophrenia
* bipolar disorder
* psychotic spectrum disorder
* lack of internet access
* lack of English fluency
* pregnant or nursing

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Use | 12 months (at baseline, 9 weeks, 3 months post-intervention, and 6 months post-intervention)
  Alcohol use will be measured using the Timeline Follow Back (TLFB) calendar. Participants will report their drinking over the past 30 days.
Change in Insomnia | 12 months (at baseline, 9 weeks, 3 months post-intervention, and 6 months post-intervention)
  Insomnia will be measured using the Insomnia Severity Index (ISI). This survey has 7 questions related to insomnia. Scores range from 0-28, with higher scores indicating increased insomnia.
Change in Sleep Quality | 12 months (at baseline, 9 weeks, 3 months post-intervention, and 6 months post-intervention)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). It measures seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Scores range from 0-indefinite. A score greater than 5 is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Weafer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University Of Kentucky Psychology Research Lab, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No